CLINICAL TRIAL: NCT03624569
Title: Cardiometabolic Benefits of Potatoes Mediated Along the Gut-Vessel Axis in Adults With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Alliance for Potato Research and Education (Other)
Responsible Party: Principal Investigator, Richard Bruno, Professor, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2018H0265
Record Dates: First submitted 2018-08-02; First posted 2018-08-10 (Actual); Results first posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Diseases; Endotoxemia; Endothelial Dysfunction; Postprandial Hyperglycemia; Gut Health
MeSH Terms: conditions — Cardiovascular Diseases; Endotoxemia; Hyperglycemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bagel diet (Sham Comparator): Bagel consumed daily for 2 weeks
  Interventions: Other: Bagel
- Potato diet (Experimental): Potato consumed daily for 2 weeks
  Interventions: Other: Potato

INTERVENTIONS:
Other: Bagel — A bagel will be consumed daily for 2 weeks.
  Arms: Bagel diet
Other: Potato — A potato will be consumed daily for 2 weeks.
  Arms: Potato diet

SUMMARY:
This study is focused on assessing potential health benefits of daily consumption of potatoes, specifically its resistant starch content (i.e. nondigestible carbohydrate), on blood vessel and gut health function in adults with metabolic syndrome. It is expected that the daily consumption of potatoes for two weeks, within a diet that follows the Dietary Guidelines for Americans, will improve blood vessel function in association with decreasing gut permeability ("leaky gut") that results in the absorption of bacterial toxins that reside in the intestine. Outcomes will therefore support dietary recommendations for potatoes to support vascular and gastrointestinal health.

DETAILED DESCRIPTION:
Cardiovascular disease is a major public health concern in the United States, where it accounts for 1 in 4 deaths every year. Vascular endothelial dysfunction is an early event leading to cardiovascular disease and can be caused by postprandial hyperglycemia. Cardiovascular disease is also characterized by metabolic endotoxemia. Metabolic endotoxemia describes increased circulating levels of gut-derived endotoxin (lipopolysaccharide; a bacterial product derived from Gram-negative bacteria in the intestines) that results from gut barrier dysfunction, a phenomenon that is common in metabolic syndrome. Studies in animals and humans have shown that consumption of resistant starch (a type of carbohydrate found in potatoes among other foods) can help to improve vascular and gut health. This clinical trial will therefore investigate the extent to which potatoes can improve microbiota composition, alleviate metabolic endotoxemia, and improve vascular function. It is hypothesized that 2-week daily ingestion of potatoes within a diet that meets the Dietary Guidelines for Americans will limit metabolic endotoxemia by decreasing gut barrier permeability and alleviating gut dysbiosis while separately improving vascular function by limiting postprandial hyperglycemia. This study will address the following objectives: 1) define changes in gut barrier function in association with improved gut microbiota composition, increased fecal short chain fatty acid (SCFA) production, and decreased serum endotoxin, 2) define changes in postprandial glycemic responses and endotoxemia, and 3) define changes in gut hormones that promote glycemic control and changes in markers of oxidative stress in relation to improvements in endothelial vascular function, all following 2-week potato consumption. To test the hypothesis, all participants will complete a randomized cross-over trial where they will receive a potato or bagel along with a diet that meets the Dietary Guidelines for Americans for 2 weeks. They will then undergo a 2-h postprandial study to define the influence of potato consumption on vascular function, glycemic control, and endotoxin translocation. Upon completing the intervention, participants will undergo a gut permeability test, fecal samples will be collected for microbiota composition analysis, and blood samples will be collected to assess endotoxin and inflammatory markers. Upon successfully completing this study, it is anticipated that chronic consumption of potatoes will be demonstrated to be an effective dietary strategy to reduce metabolic endotoxemia, improve gut health, and improve vascular function.

ELIGIBILITY:
Inclusion Criteria:

* Fasting glucose 100-125 mg/dL
* Waist circumference >102 cm (men), >88 cm (women)
* Fasting triglyceride >150 mg/dL
* Fasting HDL cholesterol <40 mg/dL (men), <50 mg/dL (women)
* Non-smoker
* Non-dietary supplement user (>1-mo)
* Free of gastrointestinal disorders, cardiovascular disease, cancer
* No recent use of antibiotics or any medications affecting glycemia, lipidemia, or blood pressure

Exclusion Criteria:

* Use of anti-inflammatory agents or probiotics
* Vegetarian, gluten-intolerant, carbohydrate-restricted diet
* Alcohol intake >2 drinks/d
* >7 hours/week of aerobic activity
* Women who are pregnant or lactating or have initiated or changed birth control in the past 3-months
* Taking medications that affect blood sugar, blood pressure, blood vessel health, or inflammation
* High blood pressure or any vascular diseases
* HIV, hepatitis, or blood disorders such as hemophilia
* Gastrointestinal disorders
* Cancer (current or past history)
* Anemia

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2020-07-16 (Actual); Study Completion 2020-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bruno, PhD, RD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data will be published as aggregate only. Data sharing may be possible pending institutional agreements.

REFERENCES:
- [Background] Cao S, Shaw EL, Quarles WR, Sasaki GY, Dey P, Hodges JK, Pokala A, Zeng M, Bruno RS. Daily Inclusion of Resistant Starch-Containing Potatoes in a Dietary Guidelines for Americans Dietary Pattern Does Not Adversely Affect Cardiometabolic Risk or Intestinal Permeability in Adults with Metabolic Syndrome: A Randomized Controlled Trial. Nutrients. 2022 Apr 8;14(8):1545. doi: 10.3390/nu14081545. PMID 35458108

RESULTS

PARTICIPANT FLOW:
Groups:
- Bagel Diet First and Potato Diet: Participants were provided a prescribed eucaloric diet for 2-weeks that contained a bagel (comparator treatment). After a washout period of 2 weeks, they then received an identical diet for 2-weeks that contained potatoes instead of bagels (comparator arm).
- Potato Diet First and Bagel Diet: Participants were provided a prescribed eucaloric diet for 2-weeks that contained a potato. After a washout period of 2 weeks, they then received an identical diet for 2-weeks that contained bagels instead of a potatoes (comparator arm).
Period: First Intervention (2 Weeks)
Arm/Group | Bagel Diet First and Potato Diet | Potato Diet First and Bagel Diet
Started | 20 | 12
Completed | 19 | 10
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2
Period: Washout (2 Weeks)
Arm/Group | Bagel Diet First and Potato Diet | Potato Diet First and Bagel Diet
Started | 19 | 10
Completed | 19 | 10
Not Completed | 0 | 0
Period: Second Intervention (2 Weeks)
Arm/Group | Bagel Diet First and Potato Diet | Potato Diet First and Bagel Diet
Started | 19 | 10
Completed | 18 | 9
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Baseline Measures - All Participants: Baseline Measures of All Participants Prior To Randomization
Arm/Group | Baseline Measures - All Participants
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 27
Body mass index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 35 (5.1)
Waist Circumference (cm) [Mean (Standard Deviation); unit: cm] | 109.8 (12.2)
Systolic Blood Pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] | 120.5 (8.4)
Diastolic Blood Pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] | 82.9 (5.6)
Plasma Glucose (mg/dl) [Mean (Standard Deviation); unit: mg/dL] | 103.7 (8.1)
Plasma High-density Lipoprotein-Cholesterol (mg/dl) [Mean (Standard Deviation); unit: mg/dL] | 36.7 (7.4)
Plasma Triglyceride (mg/dl) [Mean (Standard Deviation); unit: mg/dL] | 127.6 (80.4)
Plasma Ascorbic Acid (umol/L) [Mean (Standard Deviation); unit: umol/L] | 40.4 (21.2)

OUTCOME MEASURES:

1. Primary Outcome: Endotoxin
Description: Fasting serum endotoxin concentration
Time Frame: Day 14
Measure: Mean (Standard Deviation); unit: EU/mL
Groups:
- Bagel Diet: Participants were provided a prescribed eucaloric diet for 2-weeks that contained a bagel (comparator treatment).
- Potato Diet: Participants were provided a prescribed eucaloric diet for 2-weeks that contained a potato.
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
EU/mL | 21.2 (3.0) | 23.3 (3.0)

2. Primary Outcome: Vascular Endothelial Function
Description: Area under curve (change from baseline) for brachial artery flow-mediated dilation (FMD). The unit for FMD is %, which is calculated as: [vessel diameter in millimeters (post-occlusion) - vessel diameter in millimeters (pre-occlusion)] / vessel diameter in millimeters (pre-occlusion) x 100. FMD(%) is then used to caluclate area under the curve based on independent measures of FMD at 0-120 minutes)
Time Frame: Day 14 Postprandial (0, 30, 60, 90, 120 minutes)
Measure: Mean (Standard Error); unit: % x min
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
% x min | -259 (75) | -198 (71)

3. Secondary Outcome: Fasting Glucose Day 0
Description: Fasting plasma glucose
Time Frame: Fasting glucose on Day 0
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
mg/dL | 104 (13.5) | 109.5 (14.6)

4. Secondary Outcome: Fasting Glucose Day 14
Description: Fasting plasma glucose Day 14
Time Frame: Fasting glucose on Day 14
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
mg/dL | 101.9 (12.3) | 102.3 (13.5)

5. Secondary Outcome: Fasting Insulin Day 0
Description: Fasting plasma insulin
Time Frame: Fasting insulin on Day 0
Measure: Mean (Standard Error); unit: uIU/mL
Groups:
- Bagel Diet: Participants were provided a prescribed eucaloric diet for 2-weeks that contained a bagel part of the crossover trial (comparator treatment).
- Potato Diet: Participants were provided a prescribed eucaloric diet for 2-weeks that contained a potato part of the crossover trial.
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
uIU/mL | 21.1 (5.5) | 17.0 (2.0)

6. Secondary Outcome: Fasting Insulin Day 14
Description: Fasting plasma insulin Day 14
Time Frame: Fasting insulin on Day 14
Measure: Mean (Standard Error); unit: uIU/mL
Groups:
- Bagel Diet: Participants were provided a prescribed eucaloric diet for 2-weeks that contained a bagel (comparator treatment). part of the crossover trial
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
uIU/mL | 14.2 (2.0) | 14.9 (2.4)

7. Secondary Outcome: Postprandial Insulin
Description: Plasma insulin concentration area under curve change from baseline
Time Frame: Day 14 postprandial (0, 30, 60, 90, 120 minutes)
Measure: Mean (Standard Error); unit: uIU/mL x min
Groups:
- Bagel Diet: Participants were provided a prescribed eucaloric diet for 2-weeks that contained a bagel (comparator treatment) part of the crossover trial
- Potato Diet: Participants were provided a prescribed eucaloric diet for 2-weeks that contained a potato as part of the crossover trial.
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
uIU/mL x min | 5940 (670) | 7086 (1372)

8. Secondary Outcome: Postprandial Glucose
Description: Postprandial plasma glucose concentration area under curve change from baseline
Time Frame: Day 14 postprandial (0, 30, 60, 90, 120 minutes)
Measure: Mean (Standard Error); unit: mg/dL x min
Groups:
- Bagel Diet: Participants were provided a prescribed eucaloric diet for 2-weeks that contained a bagel as part of the crossover trial (comparator treatment).
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
mg/dL x min | 2649 (499) | 2808 (565)

9. Secondary Outcome: Fasting Endotoxin
Description: Fasting serum endotoxin concentration
Time Frame: Day 0
Measure: Mean (Standard Error); unit: EU/mL
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
EU/mL | 26.6 (2.0) | 22.3 (2.1)

10. Secondary Outcome: Postprandial Endotoxin
Description: Postprandial serum endotoxin concentration area under curve change from baseline
Time Frame: Day 14 postprandial (0, 30, 60, 90, 120 minutes)
Measure: Mean (Standard Error); unit: EU/ml x min
Groups:
- Bagel Diet: Participants were provided a prescribed eucaloric diet for 2 weeks that contained a bagel as part of the crossover trial (comparator treatment).
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
EU/ml x min | 450 (249) | -120 (176)

11. Secondary Outcome: Lactulose/Mannitol Ratio
Description: Urinary concentration of the non-digestible sugars lactulose/mannitol (mg/mg)
Time Frame: Day 14, 0-5 hours post-consumption of sugar probes
Measure: Mean (Standard Error); unit: Ratio (mg/mg)
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
Ratio (mg/mg) | .154 (.013) | .151 (0.1)

12. Secondary Outcome: Sucralose/Erythritol Ratio
Description: Urinary concentration of the non-digestible sugars sucralose/erythritol
Time Frame: Day 14, 6-24 hours post-consumption of sugar probes
Measure: Mean (Standard Error); unit: Ratio (mg/mg)
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
Ratio (mg/mg) | .0148 (0.002) | 0.01667 (0.001925)

13. Secondary Outcome: Fecal Butyrate
Description: Fecal concentration of butyrate
Time Frame: Day 14
Measure: Mean (Standard Error); unit: umol/g
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
umol/g | 21.3 (2.7) | 17.9 (2.6)

14. Secondary Outcome: Fecal Acetate
Description: Fecal concentration of acetate
Time Frame: Day 14
Measure: Mean (Standard Error); unit: umol/g
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
umol/g | 52.3 (4.7) | 46.6 (3.9)

15. Secondary Outcome: Fecal Propionate
Description: Fecal concentration of propionate
Time Frame: Day 14
Measure: Mean (Standard Error); unit: umol/g
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
umol/g | 23.1 (2.2) | 19.3 (2.1)

16. Secondary Outcome: Postprandial Cholecystokinin
Description: Plasma CCK area under curve change from baseline
Time Frame: Day 14 postprandial (0, 30, 60, 90, 120 minutes)
Measure: Mean (Standard Error); unit: pmol/L x min
Groups:
- Bagel Diet: Participants were provided a prescribed eucaloric diet for 2-weeks that contained a bagel as part of the crossover trial as part of the crossover trial (comparator treatment).
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
pmol/L x min | -196 (266) | -67 (344)

17. Secondary Outcome: Fasting Cholecystokinin
Description: Fasting plasma concentration of CCK
Time Frame: Day 14
Measure: Mean (Standard Error); unit: pmol/L
Groups:
- Bagel Diet: Participants were provided a prescribed eucaloric diet for 2-weeks that contained a bagel as part of the crossover trial.
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
pmol/L | 14.3 (3.1) | 14.2 (3.4)

18. Secondary Outcome: Postprandial NOx
Description: Plasma total nitrite/nitrate area under curve change from baseline
Time Frame: Day 14 postprandial (0, 30, 60, 90, 120 minutes)
Measure: Mean (Standard Error); unit: umol/L x min
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
umol/L x min | -240 (88) | -433 (48)

19. Secondary Outcome: Fasting NOx
Description: Fasting plasma concentration of nitrite/nitrate
Time Frame: Day 14
Measure: Mean (Standard Error); unit: umol/L x min
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
umol/L x min | 29.8 (3.7) | 30.1 (2.3)

20. Secondary Outcome: Postprandial Malondialdehyde (MDA)
Description: Plasma MDA concentration, biomarker of oxidative stress area under curve change from baseline
Time Frame: Day 14 postprandial (0, 30, 60, 90, 120 minutes)
Measure: Mean (Standard Error); unit: umol/L x min
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
umol/L x min | 57.2 (6.8) | 45.4 (7.2)

21. Secondary Outcome: Fasting Malondialdehyde (MDA)
Description: Fasting plasma MDA concentration, biomarker of oxidative stress
Time Frame: Day 14
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
umol/L | 1.78 (.1) | 1.93 (.1)

22. Secondary Outcome: Fasting Vascular Endothelial Function
Description: Fasting flow-mediated dilation of the brachial artery. Measure is calculated as: [post-occlusion vessel diameter (mm) - pre-occlusion vessel diameter (mm) / pre-occlusion vessel diameter (mm)] x 100
Time Frame: Day 14
Measure: Mean (Standard Error); unit: % change in blood vessel dilation
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
% change in blood vessel dilation | 7.2 (1.3) | 8.7 (1.3)

23. Secondary Outcome: Vitamin C
Description: Fasting vitamin C concentration, biomarker of oxidative stress
Time Frame: Day 14
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
umol/L | 47.5 (2.9) | 52.5 (4.8)

24. Secondary Outcome: cIMT
Description: Carotid intima-media thickness. Mean thickness of left and right carotid artery intima media.
Time Frame: Day 14
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
mm | 0.603 (0.109) | 0.609 (0.114)

25. Secondary Outcome: Day 14 BMI
Description: Body mass index calculated as kg weight per meters squared
Time Frame: Day 14
Measure: Mean (Standard Error); unit: kg/m^2
Groups:
- Bagel Diet: Participants were provided a prescribed eucaloric diet for 2-weeks that contained a bagel as part of the crossover trial(comparator treatment).
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
kg/m^2 | 35.1 (1.1) | 35.2 (1.1)

26. Secondary Outcome: Day 0 Waist Circumference
Description: Waist circumference in centimeters
Time Frame: Day 0
Measure: Mean (Standard Error); unit: cm
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
cm | 108.5 (2.2) | 119.1 (2.2)

27. Secondary Outcome: Day 14 Waist Circumference
Description: Waist circumference in centimeters
Time Frame: Day 14
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
mmHg | 107.8 (2.4) | 107.5 (2.4)

28. Secondary Outcome: Day 0 Diastolic Blood Pressure
Description: Diastolic blood pressure on Day 0
Time Frame: Day 0
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
mmHg | 81.5 (1.3) | 81.9 (1.5)

29. Secondary Outcome: Day 14 Diastolic Blood Pressure
Description: Diastolic blood pressure on Day 14
Time Frame: Day 14
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
mmHg | 75.9 (1.7) | 77.7 (1.4)

30. Secondary Outcome: Day 0 Systolic Blood Pressure
Description: Systolic blood pressure on Day 0
Time Frame: Day 0
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
mmHg | 123.1 (1.9) | 119.1 (2.2)

31. Secondary Outcome: Day 14 Systolic Blood Pressure
Description: Systolic blood pressure on Day 14
Time Frame: Day 14
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
mmHg | 113.6 (1.9) | 114.6 (1.8)

32. Secondary Outcome: Day 0 BMI
Description: Body mass index calculated as kg weight per meters squared
Time Frame: Day 0
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | Bagel Diet | Potato Diet
Number analyzed (Participants) | 27 | 27
kg/m^2 | 35.6 (1.2) | 35.7 (1.2)

ADVERSE EVENTS:
Time Frame: Participation in this cross-over study for each subject was approximately 8 weeks in duration.
Arm/Group | Bagel Diet | Potato Diet
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/69/NCT03624569/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/69/NCT03624569/ICF_001.pdf